CLINICAL TRIAL: NCT03902002
Title: A Single Dose, Open Label Pharmacokinetic Study of Omaveloxolone in Subjects With Mild, Moderate, or Severe Hepatic Impairment, or With Normal Hepatic Function
Brief Title: A Pharmacokinetic Study of Omaveloxolone in Subjects With Hepatic Impairment and Normal Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 408-C-1804
Record Dates: First submitted 2019-03-26; First posted 2019-04-03 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Hepatic Impairment
Keywords: RTA 408; RTA 408 capsules; Omaveloxolone; Omaveloxolone capsules; Hepatic impairment
MeSH Terms: interventions — omaveloxolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: matched healthy subjects (Experimental): On the morning of Day 1, following an overnight fast of at least 10 hours, a single oral dose of 150 mg omaveloxolone (3 × 50 mg capsules) will be administered with 240 mL of water. No food will be allowed for 4 hours post dose. Pharmacokinetic samples will be obtained from pre dose until 336 hours post dose.
  Interventions: Drug: Omaveloxolone 50 mg capsules
- Group 2: subjects with mild hepatic impairment (Experimental): On the morning of Day 1, following an overnight fast of at least 10 hours, a single oral dose of 150 mg omaveloxolone (3 × 50 mg capsules) will be administered with 240 mL of water. No food will be allowed for 4 hours post dose. Pharmacokinetic samples will be obtained from pre dose until 336 hours post dose.
  Interventions: Drug: Omaveloxolone 50 mg capsules
- Group 3: subjects with moderate hepatic impairment (Experimental): On the morning of Day 1, following an overnight fast of at least 10 hours, a single oral dose of 150 mg omaveloxolone (3 × 50 mg capsules) will be administered with 240 mL of water. No food will be allowed for 4 hours post dose. Pharmacokinetic samples will be obtained from pre dose until 336 hours post dose.
  Interventions: Drug: Omaveloxolone 50 mg capsules
- Group 4: subjects with severe hepatic impairment (Experimental): On the morning of Day 1, following an overnight fast of at least 10 hours, a single oral dose of 150 mg omaveloxolone (3 × 50 mg capsules) will be administered with 240 mL of water. No food will be allowed for 4 hours post dose. Pharmacokinetic samples will be obtained from pre dose until 336 hours post dose.
  Interventions: Drug: Omaveloxolone 50 mg capsules

INTERVENTIONS:
Drug: Omaveloxolone 50 mg capsules — Capsules containing 50 mg of omaveloxolone
  Other Names: RTA 408

SUMMARY:
This study will examine the pharmacokinetics (PK) of omaveloxolone following a single oral dose of omaveloxolone in subjects with mild, moderate, or severe hepatic impairment compared to healthy subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, of any race, between 18 and 70 years of age, inclusive.
* BMI between 18.0 and 38.0 kg/m2, inclusive, and body weight ≥ 50 kg.
* Females will not be pregnant (or planning to get pregnant) or lactating at Screening or Check in (Day 1), and females of childbearing potential and males will agree to use contraception .
* Male subjects must not donate sperm and female subjects must not donate ova from Check in (Day 1) until 90 days after their dose of study drug.

Subjects with Normal Hepatic Function Only

* Matched to subjects with mild, moderate, or severe hepatic impairment in sex, age (± 10 years), and BMI (± 20%).
* In good health, determined by no clinically significant findings from medical history, physical examination, 12 lead ECG, vital signs measurements, and clinical laboratory evaluations (congenital non hemolytic hyperbilirubinemia [e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin] is not acceptable) at Screening and Check in as assessed by the investigator (or designee).

Subjects with Hepatic Impairment Only

* Documented chronic stable liver disease (Child Pugh Class A [mild], B [moderate], or C [severe] at Screening); diagnosis of cirrhosis due to parenchymal liver disease. This will exclude biliary liver cirrhosis or other causes of hepatic impairment not related to parenchymal disorder:
* 'Documented' is defined by at least one of the following: medical history, physical examination, hepatic ultrasound, computed axial tomography scan, magnetic resonance imaging, and/or liver biopsy.
* 'Chronic stable' is defined as no clinically significant change in disease status within the last 30 days, as documented by the subject's recent medical history (e.g., no worsening of clinical signs of hepatic impairment, or no worsening of total bilirubin or prothrombin time [PT] by more than 50%).
* Subjects with mild, moderate, or severe hepatic impairment may have medical findings consistent with their hepatic dysfunction, as determined by medical history, physical examination, 12 lead ECG, vital sign measurements, and clinical laboratory evaluations at Screening and Check in (Day 1). Subjects with abnormal findings considered not clinically significant by the investigator will be eligible.

Exclusion Criteria:

* Significant history or clinical manifestation of any metabolic, allergic, dermatological, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, respiratory, endocrine, or psychiatric disorder, as determined by the investigator (or designee).
* History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the investigator (or designee).
* History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (cholecystectomy will not be allowed; uncomplicated appendectomy and hernia repair will be allowed).
* Presence of any other condition (including surgery) known to interfere with the absorption, distribution, metabolism, or excretion of medicines.
* Ventricular dysfunction or history of risk factors for Torsade de Pointes (TdP; e.g., unexplained syncope, known long QT syndrome, heart failure, and cardiomyopathy). Subjects will be excluded if there is a family history of long QT syndrome.
* Evidence of hepatorenal syndrome and estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73 m2 or abnormal sodium and potassium levels, as determined by the investigator (or designee), calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD EPI) equation at Screening or Check in (Day 1).
* Clinically significant physical examination abnormality, as determined by the investigator (or designee).
* Use or intend to use any medications/products known to alter drug absorption, metabolism, or elimination processes, including St. John's wort, within 30 days prior to dosing, unless deemed acceptable by the investigator (or designee).
* Use of any sensitive substrates for cytochrome P450 (CYP)2C8, moderate or strong inhibitors or inducers of CYP3A4/5, or substrates for p glycoprotein (P gp) within 30 days prior to study drug administration.
* Consumption of grapefruit, grapefruit products, star fruit, star fruit products, or Seville oranges within 72 hours prior to study drug administration (Day 1) and throughout the study (until after the Follow up Visit).
* History of alcoholism or drug/chemical abuse within 6 months prior to Check in (Day 1).
* Alcohol consumption of > 21 units per week for males and > 14 units for females. One unit of alcohol equals 12 oz (360 mL) beer, 1½ oz (45 mL) liquor, or 5 oz (150 mL) wine within the 6 months prior to Check in (Day 1).
* Positive urine drug screen or positive alcohol breath or urine test result at Screening and Check in (Day 1), that is not otherwise explained by permitted concomitant medications. A positive alcohol test may be repeated once at Screening. A positive alcohol test may not be repeated at Check in (Day 1).
* Positive human immunodeficiency virus test (Appendix 2).
* Participation in a clinical study involving administration of an investigational drug (new chemical entity) in the past 30 days or 10 half lives (if known), whichever is longer, prior to dosing.
* Current enrollment in another clinical study.
* Receipt of blood products within 2 months prior to Check in.
* Donation or loss of ≥ 550 mL blood from 3 months prior to Screening, plasma from 2 weeks prior to Screening, or platelets from 6 weeks prior to Screening.

Subjects with Normal Hepatic Function Only

* Confirmed supine blood pressure > 140 mmHg or < 90 mmHg and/or supine diastolic blood pressure > 90 mmHg or < 50 mmHg, or resting (supine) heart rate < 45 beats per minute (bpm) or > 100 bpm at Screening or Check in (Day 1), with a QT interval corrected for heart rate using Fridericia's method (QTcF) > 450 ms for male subjects and > 470 ms for female subjects.
* Positive hepatitis panel (Appendix 2).
* Use of tobacco or nicotine containing products within 6 months prior to Check in (Day 1), or positive cotinine at Screening or Check in (Day 1).
* Clinically significant abnormal laboratory values (clinical chemistry, hematology, coagulation, and urinalysis), as determined by the investigator (or designee).
* Significant history or clinical manifestation of hepatic disorder, as determined by the investigator (or designee).
* History or presence of liver disease or liver injury as indicated by any clinically significant deviations from normal reference ranges in liver function tests, unless approved by the investigator (or designee).
* History of diabetes mellitus.
* Use or intend to use any prescription medications/products other than prescribed hormone replacement therapy, implantable, or intrauterine contraceptives within 30 days prior to dosing, unless deemed acceptable by the investigator (or designee).
* Use or intend to use slow release medications/products considered to still be active within 30 days prior to Check in (Day 1), unless deemed acceptable by the investigator (or designee).
* Use or intend to use any non prescription medications/products including vitamins, minerals, and phytotherapeutic , herbal , or plant derived preparations within 7 days prior to Check in (Day 1), unless deemed acceptable by the investigator (or designee).

Subjects with Hepatic Impairment Only

* Confirmed supine blood pressure > 150 mmHg or < 90 mmHg and/or supine diastolic blood pressure > 90 mmHg or < 50 mmHg, or resting (supine) heart rate < 45 bpm or > 100 bpm at Screening or Check in (Day 1), with a QTcF > 470 ms for both male and female subjects.
* History of clinically significant left sided heart disease and/or clinically significant cardiac disease.
* Values outside the normal range for liver function tests that are not consistent with their hepatic condition, as determined by the investigator (or designee).
* Use of a new medication, or a change in dose, for the treatment of hepatic encephalopathy within 90 days prior to Check in (Day 1).
* Use of prescription drugs within 30 days prior to Check in (Day 1), with the exception of therapies for hepatic disease and treatment of associated disorders that had been stable for at least 3 months prior to administration of study drug (Day 1) or prescribed hormone replacement therapy, implantable, or intrauterine contraceptives.
* Recent history of, or the treatment of, esophageal bleeding (within the past 180 days), unless banded.
* History of unstable diabetes mellitus (as evidenced by hemoglobin A1c [HbA1c] ≥ 9.0% at Screening). Concomitant medications for the treatment of diabetes mellitus must be approved by the investigator (or designee), Sponsor, and Covance Medical Monitor.
* Presence of a portosystemic shunt.
* Recent history of paracentesis within 90 days prior to Check in (Day 1).
* Current functioning organ transplant or awaiting an organ transplant.
* Evidence of severe ascites.
* Recent history of hepatic encephalopathy (Grade 2 or above) within 180 days prior to Screening.
* Smoke more than 10 cigarettes or use the equivalent tobacco or nicotine containing products per day or inability to refrain from tobacco use 2 hours pre dose until 4 hours post dose.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-07-19 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of omaveloxolone in plasma | 15 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine maximum observed concentration (Cmax).
Area under the the plasma omaveloxolone concentration-time curve (AUC) | 15 days
  Pharmacokinetics will be assessed by blood sampling for omaveloxolone to determine area under the curve (AUC).

SECONDARY OUTCOMES:
Count of reported adverse events | 15 days
  Safety and tolerability will be assessed by counting adverse events, as defined the Medical Dictionary for Regulatory Activities (MedDRA).

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Orange County Research Center, Tustin, California
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/